CLINICAL TRIAL: NCT06638788
Title: Muslce Oxygenation of the Quadricep Relative to Angle and Load
Acronym: MORAL
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of British Columbia (Other)
Responsible Party: Principal Investigator, Cameron Mitchell, Assistant Professor, University of British Columbia
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: H24-01632
Record Dates: First submitted 2024-10-10; First posted 2024-10-15 (Actual); Last update posted 2024-10-15 (Actual); Status verified 2024-09

CONDITIONS: Healthy
Keywords: Muscle Oxygenation; Angle and Muscle Oxygenation; Torque and muscle oxygenation; Knee extension and muscle oxygenation

STUDY DESIGN:
Intervention Model Description: Participants will be completing loads of 20, 40, and 60% 1RM at 18,12, and 6 reps respectively on the standard knee extension (varying torque) and biodex dynamometer machine (constant torque). The muscle oxygenation of the vastus laterals muscle will be assessed throughout its range of motion in both conditions and compared to torque (standard knee extension) or knee angle (Biodex dynamometer).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Constant Torque Biodex Dynamometer (Experimental): Participants will perform their intervention on the constant torque Biodex Dynamometer
  Interventions: Other: Knee extension
- Variable Torque Standerd Knee Extension (Experimental): Participants will perform their intervention on the variable torque standerd knee extension machine
  Interventions: Other: Knee extension

INTERVENTIONS:
Other: Knee extension — Participants will perform 20, 40, and 60% of thier 1 rep maximum (1RM) at 18, 12, and 6 reps respectively.

SUMMARY:
The purpose of the present study is to determine if the amount of oxygen in muscles during resistance exercise with different weights is related to changes in torque or knee joint angle. Participants will need to come to the lab three times over three weeks. On their first visit, we will test how strong their muscles are by testing the maximal weight that can be lifted in a single repetition of a knee extension referred to as a 1 repetition maximal (1RM) followed by exercise interventions during the second and third weeks. Each exercise session will have participants lift different amounts of weight. They will use two machines: the Biodex dynamometer, that maintains constant force during a knee extension and a standard weighted knee extension machine which has variable force outputs. Participants will perform these exercises against three levels of weight, making six tests in total. Their first exercise session will take about 70 minutes and the following sessions around 55-60 minutes. They will be provided a 5-minute break between each set of lifts to ensure they are fully rested. In total, participants will be exercising for about 25-30 minutes each visit, with the rest of the time spent resting. The weights will be different percentages of the heaviest weight participants can lift.

DETAILED DESCRIPTION:
Visit 1 (70 minutes) Informed Consent and Baseline Testing Session 1

After verbal consent for participation an in-person visit will be scheduled with the associate investigator which will take place in our research space at the Chan Gunn Pavilion.

You will be asked to bring comfortable exercise clothes to this visit.

The consent form will be reviewed with you to ensure you completely understand each aspect of your involvement in the trial. If you wish to participate, you will provide written consent by signing this document in person.

Upon registration into this trial, you will complete the CSEP-Get Active Questionnaire (CSEP-GAQ), in person, which will assess your ability to safely perform exercise, as well as a general activity questionnaire to assess your exercise habits over the past 12-months. The CSEP-GAQ you complete today will be the same as the version used during your initial phone call/email screening with the study coordinator (Jacob Sanders or Ashlesh Mathrani).

Weekly physical activity will also be recorded now.

The exercise training history form will be filled out. This form will ask on average how many lower-body resistance training sets are completed per week, and on average how many minutes of lower-body moderate to vigorous physical activity are completed per week.

You will be asked to refrain from strenuous lower-body exercise for 48 hours or alcohol 12 hours before the visit, and every following visit.

We will then familiarize you with the diet and sleep forms which you will fill out at the start of every exercise intervention visit.

You will also state your dominant leg which will be used for all testing conditions

We will then randomize you to complete either variable load standard knee extensions or constant torque Biodex knee extensions in your second and third visit

You will then also be sequenced to randomly complete 20, 40, and 60% 1RM variable load standard knee extensions or constant torque Biodex knee extensions in visit 2 and 3

Upon completion of the study related forms, and randomization, height and weight will be recorded

Following these recordings, you will perform a one-repetition maximum (1RM) assessment for the knee-extension exercise on your dominant leg. This test involves slowly working up to a weight that you can move for a maximum of one full range of motion repetition.

Following the 1RM assessment, you will perform maximal isokinetic contractions on the Biodex on your dominant leg. This test involves maximum effort knee extensions at a fixed speed. This test is conducted 3 times on your dominant leg with a 2-minute rest in between tests.

Visits 2 and 3 (55/60 minutes each) Exercise Condition Visits

Visits 2 and 3 will involve a standardized warmup, filling out the sleep and diet questionnaires, and the exercise conditions in a random order. You will be asked to bring shorts and your choice of exercise top. The conditions for these visits are listed below:

Knee-extension exercises:

Dominant leg 18 repetitions at 20% 1RM set

Dominant leg 12 repetitions at 40% 1RM set

Dominant leg 6 repetitions at 60% 1RM set

Biodex exercises

Dominant leg 18 repetitions at 20% max torque set

Dominant leg 12 repetitions at 40% max torque set

Dominant leg 6 repetitions at 60% max torque set

You will arrive at the lab and will be fitted with near-infrared oxygen sensors (NIRS) on the outside of your thighs at the bottom 2/3rds between the top of the hip and the knee measuring muscle oxygenation.

You will then undergo calibration of the NIRS sensors by laying face up on a therapy table where we will then calculate your personal tourniquet pressure (PTP) on your dominant leg, a measurement used to determine pressure for a blood pressure cuff specific to your systolic blood pressure, and lower extremity limb occlusion pressure (LOP) which will determine the amount of pressure that is required for full occlusion of the arteries which will involve the cuff inflating and deflating for 20-30 seconds.

120% LOP is being used to ensure arterial flow is completely occluded. You will remain occluded until your oxygen saturation plateaus for 10 seconds (this takes between 3-5 minutes - during this time you may experience coldness/numbness in your leg and if at any point you wish to stop you can inform the research staff and the cuffs will be immediately deflated).

NIRS procedures will be performed by Jacob Sanders or Ashlesh Mathrani with specific experience and training in the procedure. These staff are not necessarily medical professionals, and it is possible that no medical professional will be in the room at the time of the procedure. Dr. Cameron Mitchell has reviewed and continues to review the performance of these procedures.

Following this plateau in saturation, the cuffs will be rapidly deflated, and you will remain face up on the therapy table until your oxygen saturation returns to resting values for two minutes.

You will then perform a general warmup on a stationary bike which will consist of 3-5 minutes of low intensity cycling at a load between 20-50W (this load will be self-selected and recorded during visit 1 and used during visits 2 and 3).

Following the general warmup you will then perform an exercise specific warmup

Six exercise tests will be performed for the variable load knee extension and constant torque Biodex knee extension split evenly with 5 minutes of rest separating sets.

Variable Load Standard Knee Extension

You will perform the knee extension exercises mentioned prior on your dominant leg and subsequently rest for 5-minutes, during which you may sit up from the leg extension machine, walk around, or use your phone/computer.

After 5 minutes of rest, you will perform the next variable load knee extension exercise test condition but this time on the dominant leg, and subsequently rest another 5 minutes.

You will repeat this procedure for the third exercise test condition as well.

All equipment used on these visits will be cleaned with disinfectant wipes before use by the next participant.

Constant Torque Biodex Dynamometer

You will perform constant torque Biodex knee extension exercises mentioned prior on your dominant leg and subsequently rest 5 minutes, during which you may sit up from the Biodex machine, walk around, or use your phone/computer.

After 5 minutes of rest, you will perform the following constant torque Biodex knee extension exercise condition and subsequently rest another 5 minutes.

After 5 minutes of rest, you will repeat the same procedure for the third exercise test condition.

All equipment used in these visits will be cleaned with disinfectant wipes following use and prior to use by the next participant.

ELIGIBILITY:
Inclusion Criteria:

1. Able to understand and communicate in English
2. All "No" answers on the CSEP Get Active questionnaire

Exclusion Criteria:

1. Current use of cigarettes or other nicotine devices
2. Any major uncontrolled cardiovascular, muscular, metabolic, and/or neurological disorders
3. Any medical condition impacting the ability to participate in maximal exercise
4. Type one or type two diabetes
5. Diagnosis of cancer or undergoing cancer treatment in the past 12 months
6. Drug therapy with any drugs that alter skeletal muscle metabolism (i.e., Metformin, Benzodiazepines, hormone replacement therapy drugs)

Ages: 19 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-09-30 (Estimated); Primary Completion 2024-11 (Estimated); Study Completion 2024-11 (Estimated)

PRIMARY OUTCOMES:
Muscle oxygenation (SmO2) curve during constant torque knee extension compared to joint angle | Within 55/60mins testing session during week 2 or 3.
  Percent of SmO2 dynamic range (%SmO2 max) will be measured during constant torque knee extension conditions at 20, 40, and 60% 1RM at 18, 12, and 6 reps respectively. The SmO2 curve for each sextile of the reps range of motion will be compared to joint angle across the three loads.
Muscle oxygenation (SmO2) curve during variable torque knee extension compared to torque | Within 55/60mins testing session during week 2 or 3.
  Percent of SmO2 dynamic range (%SmO2 max) will be measured during variable torque knee extension conditions at 20, 40, and 60% 1RM at 18, 12, and 6 reps respectively. The SmO2 curve for each sextile of the reps range of motion will be compared to torque across the three loads.

SECONDARY OUTCOMES:
Muscle oxygenation curve during variable torque compared to constant torque | Within 55/60mins testing session during week 2 or 3.
  Muscle oxygenation (%SmO2 max) curve during variable torque knee extension will be compared to the SmO2 curve during constant torque knee extension at 20, 40, 60% 1RM at 18, 12, and 6 reps respectively.

OTHER OUTCOMES:
Rate of muscle deoxygenation (%SmO2 max) compared to load for constant torque knee extension | Within 55/60mins testing session during week 2 or 3.
  Assess the rate of muscle deoxygenation (%SmO2 max) from start of set to end of set for loads of 20, 40, 60% 1RM at 18, 12, and 6 reps respectively in the constant torque condition
Rate of muscle deoxygenation (%SmO2 max) compared to load for variable torque knee extension | Within 55/60mins testing session during week 2 or 3.
  Assess the rate of muscle deoxygenation (%SmO2 max) from start of set to end of set for loads of 20, 40, 60% 1RM at 18, 12, 6 reps respectively in the variable torque condition.
Muscle oxygenation slope during eccentric compared to concentric muscle contraction in variable and constant torque knee extension | Within 55/60mins testing session during week 2 or 3.
  Muscle oxygenation (%SmO2 max) slope will be calculated for the concentric and compared to eccentric components of the knee extension range of motion at 20, 40, and 60% 1RM loads at 18, 12, and 6 reps respectively for both variable and constant torque conditions. The variable and constant torque conditions SmO2 during eccentric/concentric contractions will also be compared to each other.
Within-set muscle oxygenation slope differences during the average of the first three repetitions and the last three repetitions | 55/60 minutes in the second and third visit
  Compare within-set changes in muscle tissue oxygenation between variable load and constant load resistance exercise. Compare changes in muscle tissue reoxygenation and deoxygenation slopes averaged between first three repetitions halves and average of the last three repetitions halves of knee extension.
Muscle oxygenation (%SmO2 max) slope from minimum value to end of set during constant and variable torque knee extension | Within 55/60mins testing session during week 2 or 3.
  Muscle oxygenation (%SmO2 max) slope from minimum value to the end of set will be inspected in constant and variable torque knee extension conditions.
Minimum muscle oxygenation (SmO2) value achieved in variable and constant torque knee extension | Within 55/60mins testing session during week 2 or 3.
  Assess the minimum oxygenation value (%SmO2 max) achieved at 20, 40, and 60% 1RM at 18, 12, and 6 reps respectively during variable and constant torque knee extension repetitions.

CONTACTS AND LOCATIONS:
Overall Officials: Cameron Mitchell, B.kin, MSc, PhD, Principal Investigator — University of British Columbia

IPD SHARING:
Plan to Share IPD: Undecided